CLINICAL TRIAL: NCT01421849
Title: Patient Satisfaction and Clinical Outcomes Following Mandibular Single-implant-retained Overdenture Treatment in Residents of Nursing Homes: a Prospective Clinical Trial
Brief Title: Mandibular Single Implant Overdenture: a Prospective Clinical Trial
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Single implant in the mandible was finally not indicated due to lack of stability of the denture
Sponsor: University Hospital, Ghent (Other)
Collaborators: Southern Implants, South Africa (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2011/381
Record Dates: First submitted 2011-08-22; First posted 2011-08-23 (Estimated); Last update posted 2022-12-15 (Actual); Status verified 2022-12

CONDITIONS: Edentulous
Keywords: single implant denture; Elderly with an unstable mandibular denture
MeSH Terms: conditions — Mouth, Edentulous

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Elderly with an unstable mandibular denture. (Experimental)
  Interventions: Procedure: Denture implantation

INTERVENTIONS:
Procedure: Denture implantation — In a preliminary phase, a new denture is made according to standardized prosthodontic protocol or the old denture is adapted to provide a well-fitting denture.
  Eight weeks after insertion of the new denture an implant is placed under local anaesthetics in the centre of the mandibula.If primary stability is good, the implant is immediately loaded by the denture. If not, the implant is loaded after 6 to 12 weeks. Before, during and after the treatment patient satisfaction is evaluated by a 20 item questionnaire. Afterwards questionnaires are compared. After the insertion of the implant clinical evaluations take place at several moments.
  The total duration of the study will be 12 to 18 months.

SUMMARY:
Study hypothesis: that there would be no difference in patient satisfaction among institutionalised older people before and after treatment with a mandibular single implant-retained overdenture.

In a preliminary phase, a new denture is made or the old denture is adapted to provide a well-fitting denture.

Eight weeks after insertion of the new denture a single implant is placed in the centre of the mandibula. If the level of primary stability is sufficient to enable the implant to resist micromovement, the implant is immediately loaded . If not, the implant is loaded after 6 to 12 weeks. Primary stability is assessed by the final seating torque and by the clinician's interpretation and tactile sense of primary stability. Before, during and after the treatment patient satisfaction and clinical outcomes are evaluated by a 20 item questionnaire and a clinical examination.

ELIGIBILITY:
Inclusion Criteria:

* Edentulous residents of nursing homes treated in the mobile dental unit 'Gerodent'.
* They have to be willing to commit to 1.5 year of participation in the study.
* They have to be edentulous for at least one year before starting the implant procedure.

Exclusion Criteria:

* Medical conditions contraindicating implant surgery (unregulated diabetes type II, bisphosphonates)
* History of radiotherapy in the head and neck region
* Insufficient bone for an implant of at least 10 mm length and 4 mm diameter
* Previously treated with dental implants

Ages: 70 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-08; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Patient satisfaction after insertion of the new complete dentures. | 1 week after insertion of the new complete dentures.
  This will be measured by a questionnaire with 20 items.
Patient satisfaction after insertion of the complete dentures. | 8 weeks after insertion of the complete dentures.
  This will be measured by a questionnaire with 20 items.
Patient satisfaction post-surgical. | 1 week post-surgical.
  This will be measured by a questionnaire with 20 items.
Patient satisfaction after surgical procedure, functional loading. | 6-8 weeks after surgical procedure.
  This will be measured by a questionnaire with 20 items.
Patient satisfaction after loading the implant. | 1 week after loading the implant.
  This will be measured by a questionnaire with 20 items.
Patient satisfaction after loading. | 1 months after loading.
  This will be measured by a questionnaire with 20 items.
Patient satisfaction after loading. | 6 months after loading
  This will be measured by a questionnaire with 20 items.
Patient satisfaction after loading. | 1 year after loading
  This will be measured by a questionnaire with 20 items.

SECONDARY OUTCOMES:
Implant level : lost implants, loose implants, … | From the first week post-surgical to 1 year after loading.
Soft tissue level : Peri-implant inflammation, bleeding index, probing depth | From the first week post-surgical to 1 year after loading.
Denture related: soft tissue problems. | From 1 week after insertion of the new complete dentures to 6 months after loading.
Repair management: type (fracture, matrix replacement, patrix activation, mechanical problems of the abutment, replacement of denture, relining, adjustment without adding new material) and number. | From 8 weeks after insertion of the complete dentures to 6 months after loading.
Maintenance - oral hygiene: Implant abutment: plaque index according to Mombelli, presence of calculus. | From 1 week after loading the implant to 6 months after loading.
Maintenance - oral hygiene: Dentures using the denture plaque index by Augsburger and Elahi. | From 8 weeks after insertion of the complete dentures to 6 months after loading.

CONTACTS AND LOCATIONS:
Overall Officials: Jacques Vanobbergen, MD, PhD, Principal Investigator — University Hospital Ghent, Belgium
Locations (1):
- University Hospital Ghent, Ghent, Belgium

REFERENCES:
- See also: Related Info — http://www.uzgent.be